CLINICAL TRIAL: NCT01310998
Title: Acute Psychological Effects of High Intensity Exercise in Patients With Schizophrenia
Brief Title: Acute Psychological Effects of High Intensity Exercise With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2010/2898-3
Record Dates: First submitted 2011-01-11; First posted 2011-03-09 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; high intensity exercise; interval training exercise
MeSH Terms: conditions — Schizophrenia | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- schizophrenic disorder (Experimental)
  Interventions: Behavioral: High intensity exercise
- other psychotic disorder (Experimental)
  Interventions: Behavioral: High intensity exercise
- no mental disorder (Experimental)
  Interventions: Behavioral: High intensity exercise

INTERVENTIONS:
Behavioral: High intensity exercise — 4x4 intervals

SUMMARY:
The purpose of this study is to study the acute psychological effects in patients with schizophrenia after one session of high intensity exercise.

DETAILED DESCRIPTION:
We will examine if there is an acute effect of one high intensity session of physical exercise (4x4 intervals) on psychological variables state mood, state anxiety, well-being and psychological distress. This possible effect will be examined in three groups, one group being the main group that the other two groups will be compared up against. Group 1: Patients with schizophrenia and other psychotic illnesses. Group 2: people with non-psychotic diagnosis. Group 3: people without any psychological diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* They will be allocated into groups by their diagnoses

Exclusion Criteria:

* Not being able to complete the exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Positive and negative affects | baseline and 2 days postintervention
  Positive and Negative Affect Schedule - Expanded Form (PANSS)

SECONDARY OUTCOMES:
state anxiety | baseline and 2 days postintervention
  Questionnaire, self-report. State anxiety inventory (SAI)

CONTACTS AND LOCATIONS:
Overall Officials: Einar Vedul-Kjelsås, dr.philos, Principal Investigator — Employee at AFFU at St Olavs Hospital
Locations (1):
- Treningsklinikken, Trondheim, Norway

REFERENCES:
- [Result] Heggelund J, Kleppe KD, Morken G, Vedul-Kjelsas E. High aerobic intensity training and psychological States in patients with depression or schizophrenia. Front Psychiatry. 2014 Oct 30;5:148. doi: 10.3389/fpsyt.2014.00148. eCollection 2014. PMID 25400592